CLINICAL TRIAL: NCT06910839
Title: A PHASE 1, OPEN-LABEL, FIXED-SEQUENCE STUDY TO EVALUATE THE PHARMACOKINETIC INTERACTIONS BETWEEN PF-07976016 AND PF-06882961 IN OTHERWISE HEALTHY ADULT PARTICIPANTS WITH OVERWEIGHT OR OBESITY
Brief Title: Study to Learn About How the Study Medicines Called PF-07976016 and PF-06882961 Are Taken Up by the Body, and if Either of Them Change How the Body Processes the Other Medicine in Otherwise Healthy Adults With Overweight or Obesity
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The sponsor has made the decision to discontinue development of danuglipron (PF-06882961). As such, this study was discontinued prior to PF-06882961 administration.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C5541009
Record Dates: First submitted 2025-03-12; First posted 2025-04-04 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — danuglipron

STUDY DESIGN:
Intervention Model Description: Fixed Sequence
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Period 1 (Experimental): Participants will receive doses of PF-07976016 with and without PF-06882961
  Interventions: Drug: PF-07976016; Drug: PF-06882961

INTERVENTIONS:
Drug: PF-07976016 — PF-07976016 oral tablets
Drug: PF-06882961 — PF-06882961 oral tablets

SUMMARY:
The purpose of this study is to see how two study medicines, PF-07976016 and danuglipron, taken together affect the level of each other in the blood of participants who have overweight or obesity.

The total number of weeks of the study is up to approximately 22 weeks (5.5 months).

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant, non-breastfeeding female, 18 to 65 years of age
* BMI 25 to 40 kg/m2 and a total body weight > 50 kg (110 lb)
* Willing and able to comply with all study procedures including staying a research unit for up to 95 days

Exclusion Criteria:

* Any medical or psychiatric condition or laboratory abnormality, or recent serious illness or hospitalization, that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study including diagnosis of type 2 diabetes mellitus, type 1 or secondary forms of diabetes
* Use of any prohibited prior or concomitant medication(s)
* Presence of specified abnormalities on diagnostic assessments including clinical laboratory tests
* A positive urine drug test.
* History of alcohol abuse or repeated binge drinking and/or any other illicit drug use or dependence
* Use of tobacco/nicotine containing products in excess of the equivalent of 5 cigarettes/day or 2 chews of tobacco/day

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2025-03-13 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Steady state area under the concentration-time profile for PF-07976016 | From 0 Hours to 24 Hours following steady-state dose
Steady state maximum observed concentration (Cmax) for PF-07976016 | From 0 Hours to 24 Hours following steady-state dose
Steady state area under the concentration-time profile danuglipron | From 0 Hours to 24 Hours following steady-state dose
Steady state maximum observed concentration (Cmax) for danuglipron | From 0 Hours to 24 Hours following steady-state dose

SECONDARY OUTCOMES:
Number of participants with treatment emergent adverse events | First dose (Day 1) through 28-35 days after final dose (approximately 18 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Anaheim Clinical Trials, LLC, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5541009